CLINICAL TRIAL: NCT04757454
Title: Performance Indicators of the SARC-F Questionnaire in Acute Care
Acronym: SARC-F-CHUB
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Murielle Surquin, Head of the Internal Medicine and Geriatrics Department, Brugmann University Hospital
Other Study IDs: CHUB SARC-F
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Sarcopenia; Sensitivity; Old Age; Debility
MeSH Terms: conditions — Sarcopenia; Hypersensitivity; Frailty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 5-item SARC-F questionnaire — Administration of the 5-item SARC-F questionnaire in patients admitted to an acute care unit

SUMMARY:
The study applies the Sluggishness, Assistance in walking, Rising from a chair, Climb stairs, Falls (SARC-F) questionnaire in older patients hospitalized in an acute care geriatric unit and aims to determine its performance indicators to screen for sarcopenia according to the revised European Consensus on definition and diagnosis (EWGSOP2) within this population

DETAILED DESCRIPTION:
Sarcopenia is an age-related disease associated with health adverse outcomes, i.e. higher risk of mobility limitation, falls, fractures, mortality, and lower quality of life. The European Working Group on Sarcopenia has recently revisited one of the widely used most acknowledged definitions and launched the revised European consensus on definition and diagnosis (EWGSOP2) (4). Applying the EWGSOP2 is a three-tier process: first, screening by the Sluggishness, Assistance in walking, Rising from a chair, Climb stairs, Falls (SARC-F) questionnaire; second, diagnosis by low muscle strength, and low muscle mass; third, severity grading by low muscle function. The EWGSOP2 recommends the assessment of sarcopenia in every population, both in community-dwelling and acute care older patients. However, the evidence about the performance indicators of the SARC-F questionnaire to screen for sarcopenia in acute patients admitted to an acute care unit is really limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and over
* Hospitalized in an acute care geriatric unit due to acute health issues or acute medical conditions
* With SARC-F, hand-grip strength and dual-energy X-ray absorptiometry administered during hospital admission

Exclusion Criteria:

* SARC-F unavailable
* Unwilling to collaborate in the sarcopenia assessment
* Unwilling to sign the informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 and over hospitalized in an acute care geriatric unit due to acute medical conditions, where the SARC-F questionnaire and the EWGSOP2 was available
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the SARC-F questionnaire as screening method compared to the gold standard, which is the revised European consensus on definition and diagnosis | September 2019-November 2020
  Sensitivity, measured as a percentage (%)
Specificity of the SARC-F questionnaire as a screening method, compared to the gold standard which is the revised European Consensus on definition and diagnosis of sarcopenia (EWGSOP2) | September 2019-November 2020
  Specificity, measured as a percentage (%)
Overall concordance agreement between the SARC-F questionnaire as a screening method and the gold standard method, which is the EWGSOP2 | September 2019-November 2020
  Cohen-kappa coefficient, measured as a percentage (%)

SECONDARY OUTCOMES:
Health adverse outcomes based on the screening and diagnosis of sarcopenia as recommended by the EWGSOP2 | 1-year follow-up
  Mortality risk

CONTACTS AND LOCATIONS:
Overall Officials: Murielle Surquin, Principal Investigator — Head of the Geriatrics Department
Locations (1):
- Brugmann university hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sanchez-Rodriguez D, Marco E, Davalos-Yerovi V, Lopez-Escobar J, Messaggi-Sartor M, Barrera C, Ronquillo-Moreno N, Vazquez-Ibar O, Calle A, Inzitari M, Piotrowicz K, Duran X, Escalada F, Muniesa JM, Duarte E. Translation and Validation of the Spanish Version of the SARC-F Questionnaire to Assess Sarcopenia in Older People. J Nutr Health Aging. 2019;23(6):518-524. doi: 10.1007/s12603-019-1204-z. PMID 31233072
- [Background] Piotrowicz K, Gluszewska A, Czesak J, Fedyk-Lukasik M, Klimek E, Sanchez-Rodriguez D, Skalska A, Gryglewska B, Grodzicki T, Gasowski J. SARC-F as a case-finding tool for sarcopenia according to the EWGSOP2. National validation and comparison with other diagnostic standards. Aging Clin Exp Res. 2021 Jul;33(7):1821-1829. doi: 10.1007/s40520-020-01782-y. Epub 2021 Jan 28. PMID 33506313
- [Background] Sanchez-Rodriguez D, Marco E, Cruz-Jentoft AJ. Defining sarcopenia: some caveats and challenges. Curr Opin Clin Nutr Metab Care. 2020 Mar;23(2):127-132. doi: 10.1097/MCO.0000000000000621. PMID 31789867
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372